CLINICAL TRIAL: NCT03275077
Title: A Comparative Evaluation of Thromboelastogram and Conventional Coagulation Tests To Detect Coagulopathy in End Stage Renal Disease Patients
Brief Title: To Compare TEG (Thrombelastography) and Conventional Tests in CKD Patients
Status: Completed | Type: Observational
Sponsor: Institute of Liver and Biliary Sciences, India (Other)
Responsible Party: Principal Investigator, kelika Prakash, Asssitant Professor, Department of Anaesthesiology, Institute of Liver and Biliary Sciences, India
Other Study IDs: ILBS-TEG-001
Record Dates: First submitted 2017-08-16; First posted 2017-09-07 (Actual); Last update posted 2018-06-12 (Actual); Status verified 2018-06

CONDITIONS: End Stage Renal Disease; Coagulopathy
Keywords: End stage renal disease; ESRD; Thromboelastography; Fibrinogen
MeSH Terms: conditions — Kidney Failure, Chronic; Hemostatic Disorders | interventions — Thrombelastography

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective

GROUPS / COHORTS (2):
- Controls: Normal Healthy Volunteers
  Interventions: Device: Thromboelastography
- ESRD patients: Patients with ESRD who have not received hemodialysis. Patients with known bleeding disorders, coexisting liver diseases, those who were on antiplatelet or anticoagulant therapy and patients who had received red blood cells, fresh frozen plasma or platelet transfusions in the past three months were excluded from the study.
  Interventions: Device: Thromboelastography

INTERVENTIONS:
Device: Thromboelastography — A viscoelastic test of coagulation

SUMMARY:
Background: Coagulopathy in chronic kidney disease is multifactorial. Both hypocoagulopathy and hypercoaguability are seen. Conventional tests of coagulation (CCTs) end at the formation of thrombin, and do not take into account the interaction of coagulation factors, platelets, RBC etc. By overcoming the above deficiencies, thromboelastography provides a holistic picture of blood coagulation. The present study evaluated the TEG profile of ESRD patients and compared it to CCTs and to controls.

Methods: 50 ESRD patients and 50 controls were recruited for the study. Venous samples were withdrawn and platelet count, INR and fibrinogen levels were measured. Simultaneously a Thromboelastography was performed. All samples were drawn prior to initiation of dialysis.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy voluntary donors belonging to ASA PSI or ASA PSII
2. Patients suffering from end stage renal disease i.e. CKD stage 5 (Defined by KDIGO 2012 ) who never received renal replacement therapy (RRT)

Exclusion Criteria:

1. Patients on antiplatelet drugs, erythropoietin, desmopressin
2. Patients with known bleeding disorders like haemophilia, aplastic anaemia etc
3. Patients having coexisting liver diseases
4. Patients on dialysis
5. Patients who have received PRBC, FFPs or Platelet Transfusions in the past 3 months
6. Patients less than 18 years of age
7. Pregnant patients
8. Malignancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: A total of 100 patients were recruited for the study based on the above criteria.Following enrollment, patients were divided into two groups as follows Group 1(Control Group): 50 patients who were healthy voluntary donors belonging to ASA PSI or ASA PSII Group 2(ESRD Group): 50 patients suffering from end stage renal disease i.e. CKD stage 5 (Defined by KDIGO 2012) who never received renal replacement therapy (RRT
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2016-03-12 (Actual); Primary Completion 2016-12-22 (Actual); Study Completion 2016-12-22 (Actual)

PRIMARY OUTCOMES:
To compare the maximum amplitude on a thromboelastography in patients of chronic kidney disease stage 5 with normal controls. | 0 hr
  Maximum amplitude in whole blood will be measures by a standard kaolin thromboelastography in all patients and controls.

SECONDARY OUTCOMES:
To correlate the maximum amplitude with platelet count and fibrinogen levels in patients of chronic kidney disease | 0 hr
  the maximum amplitude obtained on an thromboelastography denotes clot strength which depends on platelet count and fibrinogen levels. thus an attempt will be made to corelate these values with fibrinogen levels and platelet count.